CLINICAL TRIAL: NCT05174247
Title: Addition of FFRct in the Diagnostic Pathway of Patients With Stable Chest Pain to Reduce Unnecessary Invasive Coronary Angiography
Brief Title: Addition of FFRct in the Diagnostic Pathway of Patients With Stable Chest Pain
Acronym: Fusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, S.P. Sharma, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MEC-2021-0189
Record Dates: First submitted 2021-11-15; First posted 2021-12-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chest Pain; Epicardial Plaques
Keywords: Stable chest pain; Coronary Angiography; major epicardial vessel stenosis
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (FFRct group) (Experimental): The people in this group receive an FFRct analysis, which will be included in the treatment plan. If the FFRct analysis shows that there are there is no significant narrowing in your case, then in principle no invasive examination (heart catheterization) performed. If the analysis indicates a significant narrowing, then an invasive cardiac catheterization will usually be required are carried out. The final treatment plan will always be reviewed by your doctor tailored to your individual situation
  Interventions: Other: FFRct analysis
- Standard treatment not using result of FFRct analyses (No Intervention): The people in this group receive the regular treatment. This is usually an invasive cardiac catheterization. The additional FFRct analysis is also included in this group, but it is not included in the treatment plan.

INTERVENTIONS:
Other: FFRct analysis — Software analysis of Cardiac CT to show extent of pericardial stenoses
  Arms: The intervention group (FFRct group)

SUMMARY:
Rationale: Patients with stable chest pain enter a diagnostic pathway where Coronary Computed Tomography Angiography (CCTA) is often the first line non-invasive test to detect coronary stenosis. An anatomically significant (≥ 50% luminal narrowing) stenosis on CCTA does however not always cause cardiac ischemia (i.e. hemodynamically significant stenosis). CCTA is often followed by invasive coronary angiography (ICA) to assess the hemodynamic significance of the stenosis which is the key determinant to decide on treatment (revascularization by coronary stenting or surgery). CCTA has a very high negative predictive value but the positive predictive value is moderate. Hence, anatomically significant stenoses on CCTA often turn out not to be hemodynamically significant on ICA. Fractional Flow Reserve from coronary computed tomography (FFRct) analysis is a new non-invasive technique that uses the CCTA images as a basis for complex software based calculations and modelling to provide additional functional information based on the anatomical CCTA images. Thus, FFRct is a totally non-invasive method. Adding the FFRct analysis to the anatomical assessment of CCTA is expected to reduce the number of patients being referred to ICA where no signs of hemodynamically significant stenosis are found on ICA.

DETAILED DESCRIPTION:
In the Netherlands, annually 180.000 new patients present with stable chest pain - the most common symptom of coronary artery disease (CAD) [1]. Stable chest pain has a 1.5% 1-year mortality and 0.7% incidence of myocardial infarction [2]. The "Kennisagenda" of the Dutch Societies of Radiology and Cardiology include CAD diagnosis as a top 10 priority.

Patients with stable chest pain enter a diagnostic pathway to detect or exclude significant coronary stenosis which is defined as > 50% luminal narrowing.

The "Verbetersignalement pijn op de borst" published by the Zorginstituut, advocates that the diagnosis should be based on a single non-invasive first line test.

Based on the National Institute for Health and Excellence (NICE) and European Society of Cardiology (ESC) guidelines, the Coronary Computed Tomography Angiography (CCTA) is a good option as the first line test in low to intermediate risk patients.

CCTA is the most sensitive non-invasive technique available, but only provides anatomical information. CCTA has an excellent negative predictive value (99%), therefore CCTA can accurately rule out CAD. However the positive predictive value is moderate (64%). Hence, anatomically significant stenoses on CCTA often turn out not to be hemodynamically significant on ICA .

Patients with significant anatomical stenosis on CCTA are often referred for invasive coronary angiography (ICA) to confirm the presence of a stenosis and subsequent revascularization of hemodynamically significant stenoses. To determine the latter, invasive fractional flow reserve (FFR) measurements can be performed during ICA. In FFR, the pressure drop across an anatomical stenosis is measured, yielding a numerical value between 0 and 1, with 1 being normal and 0.80 considered a significant stenosis.

As with all invasive procedures, ICA is associated with morbidity, mortality, patient discomfort, time and costs. Due to the moderate specificity of CCTA, many patients referred for ICA turn out to not have hemodynamically significant coronary stenosis (28-41%) in Dutch populations.

To reduce the percentage of patients referred for ICA without significant CAD, the FFRct can be useful. FFRct is a non-invasive method that uses the already acquired CCTA images to calculate coronary FFR values as they would be expected if measured invasively.

Based on data of two randomised trials conducted in the Netherlands, around 20% of patients with chest pain referred for CCTA have at least 50% anatomical coronary stenosis on CCTA . Prior FFRct studies involved populations of different countries, with different risk and work-up There are no prospective data on the real-world use of FFRct in the Dutch population of stable chest pain patients with stenosis on CCTA. The effect of FFRct in reducing unnecessary ICA or other non-invasive tests compared to CCTA alone in the Dutch health care situation is unknown. Evidence in the specific Dutch situation and population is needed to evaluate the impact and cost-effectiveness in the Dutch healthcare system.

The FUSION study is a randomized controlled trial which will investigate the impact of adding the FFRct analysis in the diagnostic pathway of stable chest pain on the rate of unnecessary ICA's.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Stable chest pain and the patient underwent CCTA which demonstrated ≥50% but less than 90% stenosis in any major epicardial vessel with a diameter ≥ 2 mm.

Exclusion Criteria:

* Inability to provide informed consent
* Unstable angina according to ESC guidelines
* Unstable clinical status
* Expected inability to complete follow-up and comply with follow-up aspects of the protocol
* History of coronary revascularisation
* Non-invasive or invasive diagnostic testing for CAD within the past 12 months (with the exception of exercise ECG)
* Unsuitable for revascularisation if required (for example due to comorbidities or anatomical features)
* Poor CT quality with expected inability to perform FFRct analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Rate of unnecessary ICA | 90 days
  Unnecessary ICA is defined as any ICA without hemodynamically significant CAD. The leading indicator for the evaluation of significant CAD is the functional measurement (FFR/iFR). If functional measurements are not available, then significant CAD is indicated by quantitative coronary angiography or ultimately by visual estimation (eyeballing).

SECONDARY OUTCOMES:
Rate of unnecessary ICA | 1 year
  Unnecessary ICA is defined as any ICA without hemodynamically significant CAD. The leading indicator for the evaluation of significant CAD is the functional measurement (FFR/iFR). If functional measurements are not available, then significant CAD is indicated by quantitative coronary angiography or ultimately by visual estimation (eyeballing).
Rate of major adverse cardiac events (MACE) | 90 days; 1 year
  Including all-cause mortality, non-fatal myocardial infarction (MI), and unplanned hospitalization leading to urgent revascularisation,
Number of additional non-invasive tests for coronary artery disease (CAD) assessment | 90 days; 1 year
Number of coronary revascularisations (planned/unplanned) | 90 days; 1 year
Rate of cardiovascular death | 90 days; 1 year
Rate of complications during and after ICA | 90 days; 1 year
Rate of non-fatal stroke | 90 days; 1 year
EuroQoL 5-Dimension 5-Level (EQ5D5L) to measure quality of life | 90 days; 1 year
  The scale used is the EQ5D5L index with a minimum value of 0 and a maximum value of 1. Higher score means that there is a higher impact on health-related quality of life.
Seattle Angina Questionnaire (SAQ) to quantify patients' symptoms of angina and the extent to which their angina affects their quality of life | 90 days; 1 year
  The SAQ is a self-report instrument with 19 items that, when scored according to the author's recommendations, yields five subscale scores: physical limitation, angina stability, angina frequency, treatment satisfaction, and disease perception. The possible range of scores for each of the five subscales is 0 to 100, with higher scores indicating better quality of life.
36-Item Short Form Survey (SF-36) to measure quality of life | 90 days; 1 year
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Cost-effectiveness | 1 year
  Calculated using the total costs (in euros) of the initial diagnostic tests, any additional tests or treatments for coronary artery disease, hospital admissions for suspected cardiac events and other costs that can be attributed to possible coronary artery disease.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo PJ Budde, MD PHD, Principal Investigator — Erasmus Medical Center; Alexander Hirsch, MD PHD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmusmc, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No